CLINICAL TRIAL: NCT06247501
Title: Treatment of CD19 Chimeric Antigen Receptor T Cells for Pediatric Patients With CD19-positive B-cell Acute Lymphoblastic Leukemia Who Are Indicated for Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-CART-CD19-SCT
Record Dates: First submitted 2024-01-17; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Very High Risk Acute Lymphoblastic Leukemia; CD19 CAR-T Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: SNUH-CD19-CAR-T — CD19 CAR-T is a gene therapy that uses genetically modified autologous peripheral blood T-cells to target CD19 on the surface of B-cells. In this approach using CARs, lymphocytes are genetically manipulated, introducing the chimeric antigen receptor gene into the lymphocytes to combine the function of effector T-cells with antibody-like abilities. The chimeric antigen receptor can recognize cell surface antigens without the need for antigen processing. By using a single-chain variable fragment (scFv) antibody, which combines the variable regions of the heavy chain (VH) and light chain (VL) through a peptide linker of approximately 15 amino acids in length, the CAR gains the ability to bind to tumor antigens.

SUMMARY:
This is a phase 2 clinical trial targeting pediatric and adolescent patients diagnosed with CD19-positive B-ALL, considered very high-risk group. The study aims to administer CD19 CAR-T therapy as an alternative to hematopoietic stem cell transplantation in patients eligible for such transplantation. The trial includes patients aged 25 or younger.

ELIGIBILITY:
Inclusion Criteria:

* Subject eligibility criteria include individuals who are under the age of 25 at the time of SNUH-CD19-CAR-T administration. Confirmation of B-cell acute lymphoblastic leukemia diagnosed at the initial assessment by a treating physician for the first diagnosis is required. Immunophenotypic analysis of CD19 expression on leukemia cells must be confirmed through immune profiling at the time of the initial diagnosis of B-cell acute lymphoblastic leukemia. In patients experiencing hematologic relapse of B-cell acute lymphoblastic leukemia, CD19 expression should also be confirmed at the time of relapse confirmation.

Patients must achieve hematologic complete remission defined as less than 5% blasts in the bone marrow after the first-line or second-line chemotherapy (first salvage therapy). Eligible patients for hematopoietic stem cell transplantation, defined by indications for transplantation, include those meeting at least one of the following criteria:

1. Philadelphia chromosome-positive due to t(9;22)(q34;q11) translocation.
2. Hypodiploidy defined by fewer than 44 chromosomes.
3. E2A-HLF gene fusion due to t(17;19) translocation.
4. Detection of minimal residual disease (MRD) positive at 0.01% or higher by next-generation sequencing confirmed after consolidation therapy and maintenance therapy.
5. Failure of the first-line therapy.
6. Cases not meeting any of the above criteria but deemed eligible for hematopoietic stem cell transplantation based on the investigator's judgment.

Exclusion Criteria:

* Patients who have undergone hematopoietic stem cell transplantation.
* Individuals for whom an adequate or sufficient leukapheresis product suitable for the production of SNUH-CD19-CAR-T cannot be obtained or is unavailable.
* Those known to be infected with the human immunodeficiency virus (HIV).
* Presence of uncontrolled active infections, determined by the investigator's assessment. If appropriate treatment has been administered for the infection, and there are no signs of progression at the time of enrollment, it is considered controlled. Persistent fever without other symptoms is not interpreted as progressive infection.
* Women who are pregnant or breastfeeding.
* Individuals deemed clinically inappropriate for participation in the clinical trial based on the investigator's clinical judgment.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival | above 3 year

SECONDARY OUTCOMES:
Overall survival | above 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea